CLINICAL TRIAL: NCT02188472
Title: PENTRIOX - a Randomized, Placebo-controlled Clinical Study on the Possible Induction of Oxidative Stress by Phenoxymethylpenicillin and Trimethoprim on Healthy Volunteers
Brief Title: Pentriox - Induction of Oxidative Stress
Acronym: PENTRIOX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henrik Enghusen Poulsen (Other)
Collaborators: Klinisk Biokemisk Afdeling (Unknown); Klinisk farmakologisk Afdeling (Unknown); Sektion for Biomedicin Institut for Veterinær Patobiologi (Unknown)
Responsible Party: Sponsor-Investigator, Henrik Enghusen Poulsen, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PEN1011
Record Dates: First submitted 2010-11-01; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Oxidative Stress
Keywords: Oxidative Stress; antibiotics
MeSH Terms: interventions — Penicillin V; Trimethoprim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Penicillin V (Active Comparator): Penicillin V 2 tablets of 330 mg twice dayly for 7 days
  Interventions: Drug: Penicillin V
- Trimethoprim (Active Comparator): 2 Tablet Trimethoprim of 100 mg twice daily for 7 days
  Interventions: Drug: Trimethoprim
- Placebo (Placebo Comparator): 2 Placebo Tablets twice daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Penicillin V — Penicillin V: 2 x 330mg tablets should be taken twice daily
  Other Names: Penicillin V, Pancillin
  Arms: Penicillin V
Drug: Trimethoprim — Trimopan: 2 x 100mg tablets should be taken twice daily
  Other Names: Trimethoprim, Trimopan
  Arms: Trimethoprim
Drug: Placebo — Placebo: 2 tablets should be taken twice daily
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate phenoxymethylpenicillin (the v-penicillin) and trimethoprim's possible induction of oxidative stress in human cells. The induction is examined by comparing changes in oxidative stress in the treatment group with the change in a placebo group. The study is a randomized-based placebo-controlled study. Each treatment group consists of 30 healthy male volunteers who consume either v-penicillins, trimethoprim or placebo over 7 days. The induction of oxidative stress is measured by 8-oxoguanosine and 8-oxodeoxoguanosine, isolated from urine. A t-test will be performed to compare drug treatment with placebo. The results will be published.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* healthy men
* non-smoker
* 18-35 years
* BMI: 18-30

Exclusion Criteria:

* Smoker
* high blood pressure
* allergies towards any of the tested medicine
* galactose-intolerance
* abnormal lipid profile
* CRP > 10
* Glucose/galactose-malabsorption
* Use of medications and herbal remedies that affect/are affected by v-penicillin and trimethoprim
* intake of narcotics 2 months prior to trial
* intake of supplements 1 month prior to trial
* bronchial asthma
* allergies
* heart deficiencies
* brady cardia
* kidney disease
* liver disease
* hypo-potassium
* phenylketonuria

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Urinary excretion of 8-oxoguanosine (nmol/24h) | Change from Baseline after seven days of treatment
Urinary excretion of 8-oxodeoxoguanosine (nmol/24h) | Change from Baseline after seven days of treatment

SECONDARY OUTCOMES:
Malondialdehyde | At the screening visit and at the final visit

CONTACTS AND LOCATIONS:
Overall Officials: Henrik E Poulsen, MD, Principal Investigator — Department head
Locations (1):
- Department of Clinical Pharmacology, Copenhagen, Denmark